CLINICAL TRIAL: NCT05501106
Title: Quality Improvement Program for the Management of Postpartum Hemorrhage After Vaginal Delivery: Protocol for A Matched-Pair, Cluster-Randomized Controlled Trial
Brief Title: Reducing Postpartum Hemorrhage After Vaginal Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Shandong Provincial Hospital (Other Government); Chongqing Medical Center for Women and Children (Other); Tianjin Central Hospital of Gynecology Obstetrics (Other); Fujian Provincial Maternity and Children's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PKUTH22-08-09
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Postpartum Hemorrhage; Vaginal Delivery
Keywords: Postpartum Hemorrhage; Vaginal Delivery; Quality Improvement
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Intervention Model Description: Recruited hospitals will be randomly assigned in a 1:1 ratio to either the experimental or comparison arms.
  All hospitals will receive general interventions, including: recommendation for implementing quality improvement programs to reduce vaginal delivery complications; trainings on obstetric quality management and clinical skills (3 times a year); and monitoring postpartum hemorrhage rate every month.
  The hospitals in the experimental group will additionally implement integrated improvement strategies which include postpartum hemorrhage risk screening, hierarchical management and preparedness, rescue recording, and case review.
Who Masked: Outcomes Assessor
Masking Description: Maternity hospital allocation will be concealed from the research assistant who will enroll and assign the hospitals. Because the quality improvement plans proposed by the NCHQMO are publicly released, it will not be possible to blind the hospital staff to the allocation. The investigators collecting information of invention implementation and acceptability will not be masked to the allocation, while the investigators assessing clinical practices and health outcomes and data statistical analysts will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison Arm (No Intervention): All hospitals will receive general interventions (comparison program), including: recommendation for implementing quality improvement programs to reduce vaginal delivery complications; trainings on obstetric quality management and clinical skills on the prediction and treatment of vaginal delivery complications (3 times a year); monitoring postpartum hemorrhage after vaginal delivery and reporting data to the NCHQMO by monitoring platform every month.
- Experimental Arm (Experimental): The hospitals in the experimental group will receive general interventions and additionally implement integrated improvement strategies which include postpartum hemorrhage risk screening, hierarchical management and preparedness, postpartum hemorrhage rescue recording, and review of postpartum hemorrhage cases (detailed in the Intervention Description).
  Interventions: Other: Integrated Improvement strategies

INTERVENTIONS:
Other: Integrated Improvement strategies — Integrated improvement strategies include postpartum hemorrhage risk screening, hierarchical management and preparedness, postpartum hemorrhage rescue recording, and review of postpartum hemorrhage cases.
  1. A checklist (named as Risk Assessment and Preparedness for Postpartum Hemorrhage (Traffic Light in Delivery Room)) will be used in each virginal delivery to help obstetric staff and teams identify risk factors after admission, before and during labor, and improve the adherence to all known best practices.
  2. The Postpartum Hemorrhage Rescue Format will be asked to be used in each postpartum hemorrhage rescue to record the rescue process.
  3. Each case of postpartum hemorrhage exceeding 1000 ml will be reviewed. We will convene a QI Panel and a Task Force to assist the hospitals in postpartum hemorrhage case review and quality improvement strategy development.
  Arms: Experimental Arm

SUMMARY:
Postpartum hemorrhage is the primary cause threatening the life safety of pregnant women in the world and China, and also the main cause of hysterectomy for women giving birth. The management of postpartum hemorrhage necessitates a coordinated multidisciplinary approach but limited available data on this issue. This program aims to evaluate the effectiveness and acceptability of the integrated strategies, on postpartum hemorrhage after vaginal delivery and relevant clinical practice, in response to the increasing incidence of postpartum hemorrhage and its long-standing threaten to the life safety of pregnant women.

A matched-pair, cluster-randomized controlled trial will be conducted among 50 maternity hospitals with at least 500 vaginal deliveries annually from five provinces in China. Recruited hospitals will be randomly assigned in a 1:1 ratio to either the experimental or comparison arms. All hospitals will receive general interventions, including: recommendation for implementing quality improvement programs to reduce vaginal delivery complications; trainings on obstetric quality management and clinical skills (3 times a year); and monitoring postpartum hemorrhage rate every month. The hospitals in the experimental group will additionally implement integrated improvement strategies which include postpartum hemorrhage risk screening, hierarchical management and preparedness, rescue recording, and case review. The primary outcome is the rate of postpartum hemorrhage, and the secondary outcomes include rate of consequent adverse outcomes, adherence to all known best practices, and staff acceptability to the interventions. These outcomes will be measured and compared between the experimental and control groups. Both intention-to-treat and per-protocol analyses will be performed.

ELIGIBILITY:
The study will be conducted at 50 hospitals in Shandong, Beijing, Tianjin, Chongqing and Fujian provinces, which are distributed in eastern and western China.

Due to the nature of the program, the unit of intervention will be at the hospital level. Hence, the recruitment plan will include selecting maternity hospitals and enrolling them into either the experimental or comparison arms.

All hospitals registered on the NCHQMO monitoring platform are required to report data of obstetric quality control indicators every month and the registration has no limitation on the hospital size, medical care level or regional distribution. The NCHQMO and the provincial centers of healthcare quality management in obstetrics in five provinces cooperate to recruit maternity hospitals from the hospitals registered on the NCHQMO monitoring platform. Each of the five provinces will contribute 10 maternity hospitals (two hospitals in each facility type: secondary public general hospitals, secondary public specialty hospitals, tertiary public general hospitals, tertiary public specialty hospitals, and private hospitals), leading to a total of 50 hospitals.

Inclusion Criteria (for hospitals):

* geographical location of the maternity hospitals within study provinces;
* being registered on the NCHQMO monitoring platform;
* willingness of the hospital leaders and staff to participate in the study;
* having at least 500 vaginal deliveries annually;
* having no potentially confounding ongoing research.

Exclusion Criteria:

-

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of postpartum hemorrhage after vaginal delivery | every month after intervention initiation
  Rate of postpartum hemorrhage after vaginal delivery (blood loss of ≥ 1000 ml within 24 hours after vaginal delivery)

SECONDARY OUTCOMES:
Rate of consequent adverse outcomes | every month after intervention initiation
  Rate of consequent adverse outcomes associated with postpartum hemorrhage, including maternal death, blood transfusion, hysterectomy, stroke, organ failure, admittance to the intensive care unit [ICU], and any other complications associated with postpartum hemorrhage.
Rate of adherence to essential clinical practices | at 6, 12, 18, and 24 months after intervention initiation
  Rate of adherence by obstetric staff to essential clinical practices for prevention and treatment of postpartum hemorrhage
Acceptability to the interventions | at 24 months after intervention initiation
  The acceptability to the interventions will be assessed through a survey among the staff from experimental hospitals at 24 months after intervention initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Yangyu Zhao, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China